CLINICAL TRIAL: NCT01212848
Title: A Pilot Safety and Feasibility Study of High Dose Left Prefrontal Transcranial Magnetic Stimulation (TMS) to Rapidly Stabilize Suicidal Patients With PTSD
Brief Title: Transcranial Magnetic Stimulation (TMS) for Suicidal Ideation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: INTRuST, Post-Traumatic Stress Disorder - Traumatic Brain Injury Clinical Consortium (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); Medical University of South Carolina (Other); Ralph H. Johnson VA Medical Center (U.S. Federal Agency); Walter Reed National Military Medical Center (U.S. Federal Agency); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INTRuST-TMS
Record Dates: First submitted 2010-09-29; First posted 2010-10-01 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Depressive Episode; Posttraumatic Stress Disorder; Traumatic Brain Injury
Keywords: Transcranial Magnetic Stimulation; Suicidal ideation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic; Suicidal Ideation | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TMS (Experimental)
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham (Sham Comparator)
  Interventions: Device: Transcranial Magnetic Stimulation - Sham Comparator

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Group 1: The treatment group will receive the following dose of repetitive TMS delivered over the left prefrontal cortex: 10 Hz, 120% Motor Threshold, 5 second pulse train, 10 second intertrain (IT) interval, 30 minutes of treatment, 6000 pulses per session; three sessions each day (18,000 stimuli) for three days for a total of 54,000 stimuli.
  Other Names: Neuronetics
  Arms: TMS
Device: Transcranial Magnetic Stimulation - Sham Comparator — The control group will receive an identical dosing schedule of "sham" repetitive TMS over three days.
  Arms: Sham

SUMMARY:
The purpose of this study is to determine whether transcranial magnetic stimulation (TMS) is effective in the treatment of suicidal thinking in individuals with a depressive episode and either posttraumatic stress disorder (PTSD), history of mild traumatic brain injury (TBI), or both conditions.

DETAILED DESCRIPTION:
Evidence suggests that depression in general, and suicidal ideation in particular, results from a dysfunctional regulatory pathway involving prefrontal cortical governance over limbic activity. Repeated daily non-invasive stimulation of the prefrontal cortex with TMS would theoretically strengthen and reset this cortical control pathway and reduce suicidal ideation and restore healthy circuit behavior.

The aim of the current study is to assess the efficacy of TMS therapy in the treatment of suicidal ideation in patients with depressive episode(s) and either PTSD or mild TBI or both. It is hypothesized that participants who receive repetitive TMS (Group 1) relative to sham treatment (Group 2) three times daily over three days will evidence more improvement in suicidal ideation from baseline to the end of day 3. Participants will be followed for six months following treatment to assess safety and long-term efficacy of TMS.

ELIGIBILITY:
Inclusion Criteria:

1. Veteran inpatients aged 18-70 years inclusive, with a depressive episode.
2. Must also have either or both

   1. a diagnosis of PTSD as defined by DSM-IV supported by the SCID, or
   2. a diagnosis of mild TBI, either complicated (i.e., with imaging abnormalities) or uncomplicated, as defined by INTRuST criteria. The American Congress of Rehabilitation Medicine (ACRM) definition of mild TBI will be utilized for this study (Kay et al., 1993). That definition will be operationalized using the INTRuST Screening Instrument.
3. Admitted because of suicidal ideation.
4. SSI score > 12.
5. HRSD question #3 > 3.
6. Female subjects of childbearing potential must have a negative urine pregnancy test.
7. Comorbid (non-principal) diagnoses of psychiatric disorders not explicitly listed in the following Exclusion Criteria section are generally permitted (with final eligibility determination by Site Principal Investigator clinical assessment).
8. Subjects must be able to speak English and complete study forms, adhere to treatment regimens, and be willing to return for regular visits.
9. After full explanation of the study, subjects must demonstrate their willingness to participate by signing the informed consent form.

Exclusion Criteria:

1. Subjects who have clinically unstable medical disease (cardiovascular, renal, gastrointestinal, pulmonary, metabolic, endocrine, other); CNS disease deemed progressive; moderate or severe traumatic brain injury (TBI). Patients with mild TBI, however, will not be excluded from study participation. The ACRM definition of mild TBI will be utilized for this study (Kay et al., 1993). That definition will be operationalized using the INTRuST TBI Screening Instrument.
2. Females who are pregnant or currently breast feeding.
3. Current or history of schizophrenia or other psychotic disorder (except psychosis NOS when the presence of sensory hallucinations are clearly related to the subject's trauma), bipolar Type I disorder, or dementia (vascular, Alzheimer's disease, other types). Patients with bipolar Type II disorder will not be excluded.
4. Subjects who repeatedly abused or were dependent upon drugs (excluding nicotine and caffeine) within 6 days of study entry will be excluded, (with the exception of alcohol abuse which, at the discretion of the primary site investigator, may be permitted*).
5. Subjects actively participating (or planning to enroll) in an evidence-based exposure/cognitive treatment for PTSD during the trial, or who have been enrolled in one during the past 6 weeks; participation in other psychotherapeutic modalities must have been stable for 3 months prior to enrollment and remain stable throughout participation.
6. Subjects currently taking medications that have short half-lives, lower the seizure threshold, and do not have evidence of antidepressant efficacy. These include high dose theophylline, or stimulants such as methylphenidate. Patients taking buproprion have to be on a stable dose and take less than or equal to 300 mg/day. Stable means the same dose for 5 half-lives.
7. Subjects with metal in their head (other than dental implants), implanted devices in their head (shunts, cochlear implants).
8. Subjects with a history of seizures or a seizure disorder.
9. Subjects with borderline personality disorder or who have clear evidence of secondary gain as a reason for admission.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-10; Primary Completion 2013-03 (Actual); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Scale of Suicidal Ideation | baseline to Day 3 of TMS treatment

SECONDARY OUTCOMES:
Safety and tolerability | baseline through 6-month follow-up.
  -adverse events, study study discontinuation due to adverse events, & decrease in cognitive function as measured by significant change on neuropsychological measures
long-term efficacy of TMS | baseline through 6-month follow-up
  -length of current hospital stay along with Scale of Suicidal Ideation score, rehospitalization rates, and suicide completion rates over 6 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Mark S George, MD, Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina

REFERENCES:
- [Derived] George MS, Raman R, Benedek DM, Pelic CG, Grammer GG, Stokes KT, Schmidt M, Spiegel C, Dealmeida N, Beaver KL, Borckardt JJ, Sun X, Jain S, Stein MB. A two-site pilot randomized 3 day trial of high dose left prefrontal repetitive transcranial magnetic stimulation (rTMS) for suicidal inpatients. Brain Stimul. 2014 May-Jun;7(3):421-31. doi: 10.1016/j.brs.2014.03.006. Epub 2014 Mar 19. PMID 24731434